CLINICAL TRIAL: NCT00458224
Title: Prevention of Permanent Obesity in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Innlandet HF (Other)
Collaborators: The Royal Norwegian Ministry of Health (Other)
Responsible Party: Principal Investigator, Trond Markestad, Professor, MD, PhD, Sykehuset Innlandet HF
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 150089
Record Dates: First submitted 2007-04-07; First posted 2007-04-10 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Overweight; Obesity; Child
Keywords: overweight; obesity; child
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Parental counseling (Experimental): Life style counseling
  Interventions: Behavioral: parental counseling

INTERVENTIONS:
Behavioral: parental counseling — Group-based family oriented program involving pediatricians, physiotherapists, dieticians, psychologists and nurses with special training
  Other Names: Life style counseling

SUMMARY:
In the county of Oppland, Norway, questionnaires addressing physical and mental health and socioeconomic status is issued to all (1960) families who meet for the pre-school assessment at the public health clinics in 2007. Particularly growth, physical activity and diet is addressed.

Families who have children with a BMI >18.9, which corresponds to BMI>30, and living in selected municipalities in the county are invited to participate in a 5 year intervention program in order to avoid future overweight conditions in children. Similarly overweight children from the rest of the county serve as controls.

DETAILED DESCRIPTION:
Background: Intervention programs to limit or reduce weight in severely obese adults and adolescents are rarely successful. In the present study intervention is aimed at moderately overweight children of 6 years.

Families in 7 municipalities who have children with BMI >18.9 are invited to a group-based family oriented program involving pediatricians, physiotherapists, dieticians, psychologists and nurses with special training. The families are invited to meet in groups times the first year, two times the second and one time the third year. According to personal interest the families are also invited to meet with the nurse between each of the the above gatherings.

The children are examined by a pediatrician before entry and after 1, 2, 3 and 5 years with specific focus on height and weight. No blood studies are routinely done.

BMI development will be related to BMIs in the family, mother's weight increase in pregnancy, socioeconomic background, general health, psychological factors scored through the Strengths And Difficulties Questionnaire, and compliance with the program. Furthermore, the results are compared to similarly overweight children from the counties who are not invited to participate in the intervention program. The results are obtained through the routine health follow-up programs in school.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 18.9
* Age 5-7 years
* Residing in Oppland county

Exclusion criteria:

* chronic disease

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2007-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Effect of BMI from a specific family oriented program | 1, 3 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Trond Markestad, Md. PhD, Principal Investigator — Sykehuset Innlandet HF
Locations (1):
- Sykehuset innlandet HF, Department of Pediatrics, Lillehammer, Norway